CLINICAL TRIAL: NCT05732753
Title: Effects of a Program Based on Mindfulness Plus Pain Neurophysiology Education Versus a Pain Neurophysiology Education Program on Perceived Quality of Life, Pain, Sleep Quality, and Functionality in Adult Patients With Non-oncological Orofacial Pain .
Brief Title: Mindfulness and Education in Patients With Non-oncological Orofacial Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jaén (Other)
Responsible Party: Principal Investigator, Agustín Aibar Almazán, Principal investigator, University of Jaén
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: -University of Jaén-
Record Dates: First submitted 2023-02-08; First posted 2023-02-17 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Oro-Facial-Digital Syndrome
MeSH Terms: conditions — Orofaciodigital Syndromes | interventions — Mindfulness; Educational Status

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: For the assignment to the groups, a random sampling will be carried out using the Epidat program. This classification will be hidden, therefore, those responsible for admitting the patients to the intervention phase will not know to which group each one has been assigned. Said assignment will be made previously by a researcher who will not intervene in the subsequent phases of evaluation, data recording intervention and database preparation. The assignment will be communicated using fully opaque sealed envelopes. The analysis of the results will be carried out by a researcher unrelated to the group assignment and the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): An experimental group (GE) that after an initial evaluation and with their consent, will be subjected to a program that includes an intervention based on Mindfulness and an 8-week Education intervention, one day a week with a duration of 120 minutes. The sessions will be divided into two parts, a part of 60' of Mindfulness and another of 60' of Education. In the Mindfulness part, formal Meditation practices and conscious movements based on yoga will be carried out. In the Education part, participants will be instructed in concepts related to the basic neurophysiology of pain.
  Interventions: Other: Mindfulness + Education in Neurophysiology of pain
- Control group (Active Comparator): The control group (CG) will receive an Education intervention, which will be evaluated in the pre and post phase of the study. Participants assigned to this group will receive 8 sessions, 60' long, with a frequency of one session per week.
  Interventions: Other: Mindfulness + Education in Neurophysiology of pain

INTERVENTIONS:
Other: Mindfulness + Education in Neurophysiology of pain — An experimental group (GE) that after an initial evaluation and with their consent, will be subjected to a program that includes an intervention based on Mindfulness and an 8-week Education intervention, one day a week with a duration of 120 minutes. The sessions will be divided into two parts, a part of 60' of Mindfulness and another of 60' of Education. In the Mindfulness part, formal Meditation practices and conscious movements based on yoga will be carried out. In the Education part, participants will be instructed in concepts related to the basic neurophysiology of pain.

SUMMARY:
To analyze the effects of a program based on Mindfulness plus Pain Neurophysiology Education versus a program based on Pain Neurophysiology Education on perceived quality of life, pain, sleep quality, and functionality, in adult patients with non-cancer orofacial pain.

DETAILED DESCRIPTION:
This research corresponds to an experimental study, a double-blind randomized controlled clinical trial, where a total of 50 men and women, over 18 years of age, will be evaluated, divided into two groups: the experimental group will receive a Mindfulness-based intervention, plus a program Education in Neurophysiology of Pain, lasting 8 weeks; and the control group will only receive an 8-week Pain Neurophysiology Education program.

The variables will be measured for both groups with the same validated tools and the same investigator to avoid information biases and differential incorrect classification. The evaluations will be carried out at the beginning of the intervention and immediately after the end of this period, and the results will be recorded in a data record that will later be unified in an Excel database, recording a code for each participant to maintain condition of privacy, but at the same time allow the required comparability.

For the independent variables, the sociodemographic characteristics will be addressed; On the other hand, the outcome variables will be the Health-Related Quality of Life [HRQOL] with the SF36 questionnaire, the Pittsburgh Index for sleep quality, the VAS scale for pain, and the Craniofacial Pain and Disability Inventory (CFPDI) for pain and functionality. Once the intervention is finished, the final evaluation will be carried out and from the comparative process define if there are significant differences with respect to the results initially obtained.

ELIGIBILITY:
Inclusion Criteria:

* Men and women older than 18 years, who voluntarily agree to participate in the study, with orofacial pain of more than 24 weeks of evolution, of non-oncological origin.

Exclusion Criteria:

* Oncological origin of orofacial pain. Systemic diseases with a focus on the TMJ. Patients operated on ATM. Population that does not agree to participate in the study or who at the time of entering the program have denied the endorsement of the use of their data for research in the informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-04-03 (Actual); Primary Completion 2023-05-29 (Actual); Study Completion 2023-06-05 (Actual)

PRIMARY OUTCOMES:
Health-related quality of life [HRQoL] with the SF36 questionnaire | Up to twelve weeks
  Used extensively for assessing health-related quality of life. For each scale, responses to each question are coded and recoded, and the results are transferred to a 0-100 point scale. On this scale of 0-100 of the SF-36, the higher the score obtained, the better the state of health.
Pain with VAS scale | Up to twelve weeks
  Scale used to help a person rate the intensity of certain sensations and feelings, such as pain. Depending on the cm indicated by the patient, the value of said self-report is extrapolated to a numerical value that will be: no pain=0; mild pain=1.2; moderate=3-5; intense=6-8; unbearable=9-10.
Pain and functionality with Craniofacial Pain and Disability Inventory (CF-PDI) | Up to twelve weeks
  Questionnaire composed of 21 items, allows to improve the diagnosis in patients with primary and secondary headaches, and in those with temporomandibular disorders or some other orofacial pain.
Quality of sleep with the Pittsburgh Index | Up to twelve weeks
  A simple and valid assessment of both sleep quality and disturbance that might affect sleep quality.

CONTACTS AND LOCATIONS:
Locations (1):
- Maxillofacial Surgery service of the Hospitals: Virgen de las Nieves of Granada and Neurotraumatology of Jaén., Jaén, Spain

IPD SHARING:
Plan to Share IPD: No